CLINICAL TRIAL: NCT02922387
Title: Varenicline and Advanced Behavioral Support on Smoking Cessation and Quality of Life in Inpatients With Acute Exacerbation of COPD, Bronchial Asthma Attack, or Community-acquired Pneumonia: a Prospective Open-label 52-week Follow-up Trial
Brief Title: Smoking Cessation Intervention in Respiratory Inpatients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General Hospital of Kavala (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, ALEXIOS POLITIS, Principal Investigator, General Hospital of Kavala
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTBSQOL-52-CAC
Record Dates: First submitted 2016-09-27; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma; Community Acquired Pneumonia
Keywords: varenicline; COPD; asthma; pneumonia; smoking cessation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Community-Acquired Pneumonia; Pneumonia; Smoking Cessation | interventions — Varenicline; Behavior Therapy; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline + Behavioral support (Experimental): varenicline and behavioral support
  Interventions: Drug: Varenicline; Behavioral: Behavioral support
- Behavioral support (Active Comparator): behavioral support
  Interventions: Behavioral: Behavioral support

INTERVENTIONS:
Drug: Varenicline — Varenicline was given for 12 weeks to all patients in group A. The initial dose was 0.5 mg/day for days 1-3, and was then up-titrated to 0.5mg on days 4-7, and finally to 1 mg twice daily from day 8 until the end of treatment
  Other Names: Chantix
  Arms: Varenicline + Behavioral support
Behavioral: Behavioral support — An initial private consultation session and motivational interview while still in the hospital that lasted for at least 60 minutes. Follow-up phone calls with a minimum duration of 10 minutes were scheduled in weeks 1, 2, 4, and months 3,6 and 9 following smoking cessation.
  Other Names: motivational interview; consultation session

SUMMARY:
Prospective, open-label, parallel-group, 52-week trial comparing varenicline in combination with behavioral support with one session of behavioral support alone.

Eligible patients were smokers hospitalized due to a) acute exacerbation of chronic obstructive pulmonary disease (COPD), or b) bronchial asthma attack, or c) community-acquired pneumonia (CAP).

The primary outcome was the success rate (%) at week 52. Secondary outcomes were quality of life (QoL) alterations on the domains of the 36-Item Short Form Health Survey (SF36) and investigation of possible predictors for smoking abstinence.

DETAILED DESCRIPTION:
Patients screened for eligibility were all the smokers who were hospitalized in the First Pulmonology Clinic of Kavala General Hospital from May 2012 to May 2014.

Patients had an initial private consultation session and motivational interview while still in the hospital. Following this interview, patients chose the smoking cessation intervention they preferred: either the standard regimen for varenicline and behavioral support or behavioral support without pharmacotherapy.

All patients quit smoking while still hospitalized.Follow-up phone calls with a minimum duration of 10 minutes were scheduled in weeks 1, 2, 4, and months 3,6 and 9 following smoking cessation.

Patients in both groups were asked to return to hospital in month 12 (week 52) for a final assessment. At this last visit, the SF36 was again completed and exhaled CO was (re) measured.

ELIGIBILITY:
Inclusion criteria:

* Adult smokers (> 100 cigarettes in their lifetime)
* Patients hospitalized due to either a) acute exacerbation of COPD, or b) acute exacerbation of bronchial asthma, or c) community acquired pneumonia.
* Patients who agreed to participate and provided written informed consent were recruited.

Exclusion criteria:

* Inpatients younger than 18
* adult smokers hospitalized for any reason other than acute exacerbation of COPD / bronchial asthma or community acquired pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation Rate at week 52 | 12 months follow up

SECONDARY OUTCOMES:
Quality of life changes following smoking cessation | 12 months follow up
  Quality of life (QoL) was assessed, in both groups, with the Short Form SF36 questionnaire at baseline and at the end of the followup period, week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos I Gourgoulianis, Prof., Study Director — Department of Respiratory Medicine, Faculty of Medicine, School of Health Sciences, University of Thessaly, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No